CLINICAL TRIAL: NCT04105907
Title: Histological Evaluation in the Efficacy of GentleWave in Root Canal Pulp Tissue Debridement and Disinfection of Difficult to Reach Areas in Mandibular Human Molars II. An In-vivo Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Sonendo, Inc. (Industry)
Responsible Party: Principal Investigator, David E Jaramillo, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-19-0476
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Root Canal Treatment
Keywords: GentleWave; Multisonication; Sonendo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Partial root canal treatment with the Sonendo GentleWave (Experimental)
  Interventions: Device: GentleWave

INTERVENTIONS:
Device: GentleWave — Subject teeth will receive a partial root canal treatment with the Sonendo GentleWave system followed by extraction of the tooth and histological evaluation of the tooth

SUMMARY:
The purpose of this study is to understand and learn better the efficacy of GentleWave and obtain histological evidence of the efficacy of this new technology done in-vivo

ELIGIBILITY:
Inclusion Criteria:

* Only teeth that patient decided to have the extraction done instead of having any other type of dental treatment and teeth extracted at patient's petition.

Exclusion Criteria:

* Teeth with root fractures or previously root canal treated teeth.
* Teeth with severe loss of structure
* Children

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Visualization of the amount of pulp tissue left behind after GentleWave procedure | at the time of tooth extraction(immediately after GentleWave procedure)
  Visualization of the amount of pulp tissue left behind after GentleWave procedure as assessed by reviewing the histological serial sections under the light microscope

SECONDARY OUTCOMES:
Number of participants with the presence of bacteria inside the root canal and inside the dentinal tubules as assessed by observation under the light microscope | at the time of tooth extraction(immediately after GentleWave procedure)

CONTACTS AND LOCATIONS:
Overall Officials: David E Jaramillo, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No